CLINICAL TRIAL: NCT00992290
Title: Probiotic LGG in Patients With Minimal Hepatic Encephalopathy
Brief Title: Probiotic Lactobacillus GG (LGG) in Patients With Minimal Hepatic Encephalopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM12123; 1U01AT004428-01A1 (NIH)
Record Dates: First submitted 2009-10-06; First posted 2009-10-09 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Minimal Hepatic Encephalopathy
Keywords: cirrhosis; hepatic encephalopathy; complications; probiotic; lactobacillus GG
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus GG (Experimental)
  Interventions: Biological: Lactobacillus GG
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Lactobacillus GG — 1 capsule of lactobacillus GG BID compared to placebo BID
  Arms: Lactobacillus GG
Biological: Placebo — 1 capsule of lactobacillus GG BID compared to placebo BID
  Arms: Placebo

SUMMARY:
This research proposes to find whether the probiotic lactobacillus GG is safe and well tolerated in patients with minimal hepatic encephalopathy. We also want to get insight into the mechanisms of action of LGG.

DETAILED DESCRIPTION:
Development of complementary and alternative medicine approaches to liver disease is a priority area at NCCAM. Minimal hepatic encephalopathy (MHE) is a significant complication of cirrhosis which can result in poor quality of life, impaired cognition and difficulty in driving motor vehicles with a high traffic accident risk. MHE is estimated to affect one half of the 5.5 million cirrhotics in the U.S. Despite these negative outcomes, there is no consensus on treatment of MHE. Currently available therapies for MHE act on intestinal flora but are limited by adverse effects (i.e. lactulose-induced diarrhea), which negatively impact adherence. Probiotic bacterial supplements, which also act on intestinal flora, are an emerging therapy for MHE. Our group has performed a pilot, randomized trial which demonstrated a significantly higher rate of MHE reversal with excellent adherence in patients randomized to probiotic yogurt compared to no therapy. This proposal intends to define Lactobacillus GG (LGG) as a biologically-based alternative therapy for MHE with special focus on metabolic and stool bacteriologic changes.

The hypothesis of this Phase I proposal is: LGG will be safe and efficacious for the treatment of minimal hepatic encephalopathy compared to placebo in a randomized, double-blind trial.

This will be carried out with four specific aims:

Specific aim 1: To define the safety and tolerability of LGG in patients with minimal hepatic encephalopathy against placebo in a Phase I randomized controlled trial.

Specific aim 2: To define the effect of LGG on intestinal microflora composition in cirrhotics with minimal hepatic encephalopathy using 16s stool DNA sequencing in a randomized, placebo-controlled trial.

Specific aim 3: To determine the effect of LGG on metabolic biomarkers and cytokines in stool, urine and blood using nuclear magnetic resonance spectroscopy in minimal hepatic encephalopathy.

Specific aim 4: To determine the effect of LGG on psychometric function in patients with minimal hepatic encephalopathy.

The specific aim and sub-aims will be tested in 30 patients with non-alcoholic cirrhosis and MHE: 15 randomized to LGG and 15 randomized to placebo to be taken BID for 8 weeks with detailed psychometric, metabolic, anthropometric and bacteriologic evaluation. Results generated from this study will form the basis for a RO1 proposal to develop the use of probiotics as a biologically-based alternative treatment with long-term outcomes of prognosis, development of overt encephalopathy and prevention of traffic accidents in patients with MHE.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* Histological evidence of cirrhosis
* Maintenance of cirrhosis treatment and stability for 6 months
* Mini-mental state exam score > 25
* Presence of MHE on psychometric testing

Exclusion Criteria:

* Rx for MHE or OHE
* Antibiotics within 6 weeks
* Yogurt consumption within 2 weeks
* Neutrophil count < 500
* Inflammatory bowel disease
* History of pancreatitis
* Hepato-cellular carcinoma
* Recent (6 weeks) gastrointestinal bleed
* Recent (6 months) alcohol intake
* Psychoactive medications (including interferon/antipsychotics)
* Liver transplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-10; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety of LGG | 3 years

SECONDARY OUTCOMES:
Quality of life measured by sickness impact profile | 3 years
Bacteriology measured in the stool flora by specialized non-culture techniques | 3 years
Metabonomics and psychometric testing using a standard psychometric battery | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan S Bajaj, MD, MSc, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States